CLINICAL TRIAL: NCT01555606
Title: A Multicenter, Observational, Noninterventional, Narrative Study to Evaluate Patient-Reported Experiences of Living With Moderate-to-Severe Plaque Psoriasis
Brief Title: An Observational Study to Evaluate Patient-Reported Experiences of Living With Moderate-to-Severe Plaque Psoriasis
Status: Completed | Type: Observational
Sponsor: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100687; NOCOMPOUNDPSO4001 (Other: Janssen Biotech)
Record Dates: First submitted 2012-03-14; First posted 2012-03-15 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: Psoriasis; Patient-reported outcome; Quality of Life
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Moderate to severe plaque psoriasis patients: The group includes adult patients (either male or female) diagnosed with plaque psoriasis for at least 6 months prior to screening with PGA value of greater than or equal to 3. The patients in the group needed are currently receiving treatment with conventional systemic agents, topical therapy and/or phototherapy or biologic therapy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Patients will not be administered any treatment as part of the study and will receive usual care. Patients will be evaluated for PROs by obtaining narratives and photographs.

SUMMARY:
The purpose of the study is to develop a database containing patient-reported information that may be used to understand and to increase awareness of the impact that moderate-to-severe plaque psoriasis can have on both daily life and life in general from a patient's perspective. The database will include self-reported patient narratives on the topic of the experience of having moderate-to-severe plaque psoriasis and will include information on treatments received, as well as de-identified clinical photographs taken over the course of the disease.

DETAILED DESCRIPTION:
This study is planned with the primary objective of developing a database containing patient-reported information that may be used to understand and increase awareness of the impact that moderate-to-severe plaque psoriasis can have on both daily life and life in general from a patient's perspective. This is a multicenter observational (no drug given to the patient) patient narrative study. The duration of study is 16 weeks and includes adult patients with moderate-to-severe plaque psoriasis who are candidates for phototherapy or systemic therapy. The study investigators are dermatologists who treat patients with moderate-to-severe plaque psoriasis. The study includes a screening visit 2 weeks before Week 0 (baseline). Patients will be evaluated at screening for current or peak historical physician's global assessment (PGA) response (range 0-5). Patients will provide narratives at the Week 0 (baseline) visit and may add additional information at an interval visit or at the end of the study on Week 16. Photography will be performed at Week 0 and at the end of study at Week 16. Additional photographs will be taken if there is any change in disease status (e.g., disease improvement or worsening, change in treatment) occurring prior to the end of the study. Between Week 0 and Week 16, patients may return to the study site for 1 interval visit at the first clinically significant change in disease status, if applicable. The Week 16 final assessment may be conducted as a telephone follow-up for patients who have had an interval visit between Week 0 and Week 16. If the patient did not return to the study site for an interval visit, the patient will return to the study site for a visit at Week 16. All assessments specified for the interval visit will be performed at Week 16. All patients will have the following data collected: PGA score, area of body involved, body surface area percent (BSA%, calculates percent of body surface area affected with psoriasis), Psoriasis Area and Severity Index (PASI) de-identified photographs, adverse events, and patient narratives. The information will be collected de-identified. Study materials (e.g., demographic and disease characteristic forms, narratives, and photographs) will be coded using a unique patient identification (ID) number. Only de-identified information will be available to the Sponsor and related study personnel.

ELIGIBILITY:
Inclusion Criteria:

Adult male and female patients having diagnosis of plaque psoriasis for at least 6 months prior to screening

* Patients who are candidates for or are currently receiving the following: a. conventional systemic agents (eg, MTX, acitretin, cyclosporine, fumarates, or systemic psoralens plus ultraviolet A light [PUVA]), b. topical therapy and/or phototherapy (and are eligible for, but are not currently receiving oral systemic or biologic therapy), c. biologic therapy for moderate to severe plaque psoriasis
* Have a peak historical or current physician's global assessment (PGA) of greater than or equal to 3 (range 0-5)
* Patients must have the ability to read and speak English
* Patients must reside in the US.

Exclusion Criteria:

Patients with guttate, erythrodermic, or pustular psoriasis (all are various types of psoriasis)

- Patients with serious concomitant illness that could require the use of systemic corticosteroids or otherwise interfere with the patient's participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes adult patients with moderate-to-severe plaque psoriasis who are candidates for phototherapy or systemic therapy
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To develop a database for patients with moderate-to-severe plaque psoriasis containing patient-reported information | Week 0 to Week 16
  The database will contain patient-reported information that may be used to understand and increase awareness of the impact that moderate-to-severe plaque psoriasis can have on both daily life and life in general from a patient's perspective. The database will include self-reported patient narratives on the topic of the experience of having moderate-to-severe plaque psoriasis, information on treatments received, and de-identified clinical photographs taken over the course of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Biotech, Inc. Clinical Trial, Study Director — Janssen Biotech, Inc.
Locations (9):
- United States (9):
  - Phoenix, Arizona
  - Sacramento, California
  - Ann Arbor, Michigan
  - East Windsor, New Jersey
  - Stony Brook, New York
  - Winston-Salem, North Carolina
  - Murfreesboro, Tennessee
  - Dallas, Texas
  - Norfolk, Virginia

REFERENCES:
- [Result] Pariser D, Schenkel B, Carter C, Farahi K, Brown TM, Ellis CN; Psoriasis Patient Interview Study Group. A multicenter, non-interventional study to evaluate patient-reported experiences of living with psoriasis. J Dermatolog Treat. 2016;27(1):19-26. doi: 10.3109/09546634.2015.1044492. Epub 2015 Jul 3. PMID 26138406